CLINICAL TRIAL: NCT05829304
Title: A Comparative Clinical and Radiographic Study Of Collagen Based Pulpotomy Versus MTA Pulpotomy in Cariously Exposed Vital Primary Molars
Brief Title: A Comparative Clinical and Radiographic Study Of Collagen Based Pulpotomy in Cariously Exposed Vital Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: sherouk atef elsayed (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, sherouk atef elsayed, A comparative Clinical and Radiographic Study Of Collagen based Pulpotomy Versus MTA Pulpotomy in Cariously Exposed Vital Primary Molars, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 251293
Record Dates: First submitted 2022-12-21; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Dental Caries in Children

STUDY DESIGN:
Intervention Model Description: Teeth that will be included in the current trial will be randomly assigned one of the experimental groups using closed white envelopes (simple randomization 1:1 ratio).
Who Masked: Participant, Outcomes Assessor
Masking Description: the blinding is not possible (unfortunately) due to the nature of the trial. Trial participants, outcome assessors and statistician will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen based pulpotomy (Active Comparator): Application of rubber dam for isolation, then a standardized pulpotomy procedure will be performed. Remove pulpal tissues to the orifice level. Haemostasis will be achieved by the application of a wet cotton pellet.
  Group I collagen-based Pulpotomy:
  1. After complete haemostasis, collagen based pulpotomy will be applied according to the manufacturer's instructions and gently placed over the pulp stumps to a thickness of 2 mm then the rest of the pulp chamber will be filled with glass ionomer cement.
  2. Tooth will be restored with stainless steel crown.
  Interventions: Other: MTA based pulpotomy; Other: Collagen based pulpotomy
- MTA based pulpotomy (Active Comparator): Application of rubber dam for isolation, then a standardized pulpotomy procedure will be performed. Remove pulpal tissues to the orifice level. Haemostasis will be achieved by the application of a wet cotton pellet.
  Group II MTA pulpotomy:
  1. After complete hemostasis, MTA+ Cerkamed will be manipulated to obtain a putty mix. This mix will be placed over the radicular pulp. condensation of the mix with a moistened cotton pellet, followed by application of glass ionomer cement.
  2. Tooth will then be restored with stainless steel crown.
  Interventions: Other: MTA based pulpotomy; Other: Collagen based pulpotomy

INTERVENTIONS:
Other: MTA based pulpotomy — The principal investigator will carry out all treatment procedures, and the patients will be assigned. It will be as split mouth, both groups A&B will be at the same patient.
Other: Collagen based pulpotomy — The principal investigator will carry out all treatment procedures, and the patients will be assigned. It will be as split mouth, both groups A&B will be at the same patient.

SUMMARY:
To assess post operative pain and survival rate after collagen based pulpotomy versus MTA pulpotomy in children with vital primary molars.

DETAILED DESCRIPTION:
Pulpotomy of vital primary molars is indicated when caries removal results in pulp exposure. Treatment approaches consist of devitalization using formocresol, preservation using ferric sulfate and regeneration using mineral trioxide aggregate of the remaining pulp tissue have been utilized to date. The ideal pulpotomy medicament would be biocompatible and bactericidal, in addition, to promote the healing of the root pulp and be compatible with the physiological process of root resorption.

Collagen, which is available for dental implication, is already sterilized and also reinforced with antibiotic particles to efficiently aid in regeneration and repair without any contaminations. The collagen particles can be sterilized by various methods like irradiation, dry heat, and ethylene oxide, among which irradiation is the most frequently used method as it does not affect the structural stability

ELIGIBILITY:
Inclusion Criteria:

1. Primary molar tooth not more than one-third of root resorption.
2. Children with bilateral deep dental caries approximating the pulp in primary molars assessed both clinically and radiographically.
3. systemically healthy.
4. cooperative patients who will comply to follow up visits.

Exclusion Criteria:

1. Children with medical, physical, or mental conditions.
2. Primary molars with any congenital deformities.
3. Previously accessed teeth.
4. At operative procedure haemorrhage control is unachievable after pulpotomy.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 19 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | 3 days
  postoperative pain following the placement of restoration by questioning the patient. using numerical pain rating scale Zero means patient have no pain, while 10 represents the most intense pain possible.

SECONDARY OUTCOMES:
Absence of internal root resorption | up to 24 week
  binary outcome detected with periapical x-ray by parallel technique using XCP film holder
absence of swelling | up to 24 week
  binary outcome detected with periapical x-ray by parallel technique using XCP film holder

REFERENCES:
- [Background] Anandan V, Inbanathan J, Saket P, Krishnamoorthy V, Gandhi S, Chandrababu VK. Assessment of Clinical and Radiographic Success Rate of Formocresol-based Pulpotomy versus Collagen-based Pulpotomy: An In Vivo Study. J Contemp Dent Pract. 2021 Jun 1;22(6):680-685. PMID 34393127